CLINICAL TRIAL: NCT01852097
Title: A Pilot Randomised Controlled Trial to Determine the Feasibility, Acceptability and Effectiveness of a CBT Based Online Intervention to Address Practical and Perceptual Barriers to Medication Adherence in Inflammatory Bowel Disease.
Brief Title: An Online Intervention to Address Barriers to IBD Medication Adherence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12/0210
Record Dates: First submitted 2012-10-11; First posted 2013-05-13 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-02

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Inflammatory Bowel Disease (IBD); Crohn's disease; Ulcerative colitis; Cognitive Behavioural Therapy (CBT); Medication adherence
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT based online intervention (Experimental): CBT based online intervention to elicit and address perceptual and practical barriers to taking medication.
  Interventions: Behavioral: CBT based online intervention to elicit and address perceptual and practical barriers to taking medication.
- Control group (No Intervention): Care as Usual. Participants in the control group will be able to access the online intervention after they complete their last follow-up questionnaire.

INTERVENTIONS:
Behavioral: CBT based online intervention to elicit and address perceptual and practical barriers to taking medication. — The general approach to the intervention is the following:
  1. Assess and profile individual perceptual and practical barriers to medication for IBD using validated questionnaires.
  2. Give feedback to individuals on their questionnaire responses.
  3. Provide individualised advice to address doubts, misconceptions and concerns for currently prescribed medications.
  4. Provide advice on overcoming practical barriers.
  5. Send motivational messages (and reminders if applicable) by email or text based on the unique profile of each participant.
  6. Provide information about how to raise concerns with medical practitioners and how to get the most from a medical consultation.
  Arms: CBT based online intervention

SUMMARY:
Background Inflammatory Bowel Disease (IBD) is a group of lifelong and relapsing inflammatory conditions that usually affect the colon and the small intestine. Between 30 to 45% of patients with IBD do not take their treatment as prescribed by their health care team (Jackson, Clatworthy et al. 2010). The Perceptions and Practicalities Approach (PAPA) provides a theoretical framework to develop adherence interventions that are patient-centred (Horne, 2001). Unintentional non-adherence occurs when the patient wants to take the medication but there are barriers beyond their control, such as not understanding the instructions (practical barriers). Intentional non-adherence is the result of the beliefs affecting the patient's motivation to continue with treatment (perceptual barriers).

Aims

1. To develop an internet-based intervention to address perceptual and practical barriers to adherence to medicine for IBD.
2. To determine whether the intervention is effective based on change in both types of barriers.

Plan of Investigation The inclusion criteria are: age 18 or over; diagnosis of IBD; currently prescribed azathioprine, mesalazine, and/or adalimumab.

240 participants identified via Crohn's and Colitis UK and through two NHS IBD clinics will take part in the study. An online pilot Randomised Controlled Trial will allocate the participants either to a Cognitive Behavioural Therapy (CBT) based online intervention or Treatment as Usual group. On first visiting the website, participants will be screened for eligibility and asked for consent before answering the questionnaires. The website will assign intervention modules to be completed based on an individual's profile.

Outcomes: Beliefs about Medicines scores will be measured at baseline, 1 month and 3 month follow-ups.

Potential Impact A CBT based online intervention tailored to personal needs and concerns may benefit a large number of patients with low costs for the national healthcare services. A website can be accessed at a time and place convenient to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over.
* Diagnosis of IBD (Crohn's Disease or Ulcerative Colitis or Indeterminate Colitis).
* Currently prescribed one or more of the following medications for IBD: azathioprine, mesalazine, and adalimumab.

Exclusion Criteria:

* We will exclude people who are for any reason unable to make an informed decision about taking part and people who do not wish to complete follow-up questionnaires.
* People who declare that they do not understand written English. This is a pilot feasibility study that aims to assess the effectiveness and acceptability of an online CBT based intervention in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-11 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Change in Beliefs about Medicines Questionnaire (BMQ) | Baseline, 1 month follow-up, 3 month follow-up
  The BMQ (Horne and Weinman, 1999) has been validated for use with people with chronic conditions. It comprises a scale that measures beliefs about medication prescribed specifically for IBD and a general scale that evaluates beliefs that medicines are harmful, addictive, poisons.

SECONDARY OUTCOMES:
Change in Medication Adherence Report Scale (MARS) | Baseline, 1 month follow-up, 3 month follow-up
  The MARS scale (Horne and Hankins 1997) is extensively used as a measure of adherent behaviours in a variant of illness populations. The MARS attempts to diminish the social pressure on patients to under-report non-adherence by phrasing adherence questions in a non-threatening manner and assuring them that responses are anonymous and confidential.
Change in Hospital Anxiety and Depression questionnaire (HADS) | Baseline, 1 month follow-up, 3 month follow-up
  The HADS scale (Zigmond and Snaith 1983) is a reliable and valid instrument for detecting states of depression and anxiety.
Change in Visual Analogue measure of adherence | Baseline, 1 month follow-up, 3 month follow-up.
  Self-reported estimation of the % of medication taken over the last 4 weeks.
Change in Brief Illness Perception Questionnaire (IPQ) | Baseline, 1 month follow-up, 3 month follow-up.
  The brief IPQ (Broadbent, Petrie et al. 2006) has demonstrated adequate test-retest reliability and validity.
Change in Satisfaction with Information about Medicines Scale (SIMS) | Baseline, 1 month follow-up, 3 month follow-up
  The SIMS scale (Horne, Hankins et al. 2001) is a valid and reliable instrument for assessing how well the needs for medicines information in patient are being covered.
Change in Marlow-Crowne Social Desirability Scale-Form C (M-C Form C) (Reynolds 1982) | Baseline, 1 month follow-up, 3 month follow-up
  The Marlow-Crowne Social Desirability Scale-Form C (Reynolds 1982) is a measure of social desirability as a response tendency and it has been proved reliable and consistent (Nordholm 1974; Crino, Rubenfeld et al. 1985; Barger 2002).
Change in Short Inflammatory Bowel Disease Questionnaire | Baseline, 1 month follow-up, 3 month follow-up
  The SIBDQ is a valid and reliable tool able to detect meaningful clinical changes in the health related quality of life of individuals with both Crohn's disease and Ulcerative colitis. It measures physical, social, and emotional status (the scores go from 10 to 70, poor to good quality of life).

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- See also: Sponsor — http://www.ucl.ac.uk/jro
- See also: UCL School of Pharmacy official website — http://www.ucl.ac.uk/pharmacy